CLINICAL TRIAL: NCT06115642
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Characteristics of HLX43 (Anti-PD-L1 ADC) in Patients With Advanced/Metastatic Solid Tumors
Brief Title: A Phase I Study to Evaluate the Safety, Tolerability, and PK of HLX43 in Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX43-FIH101
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Advanced/Metastatic Malignant Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Ia (Dose Escalation) (Experimental): Patients with advanced/metastatic solid tumors
  Interventions: Drug: HLX43
- NSCLC failed to standard treatment (Part 2 Dose Expansion) (Experimental): Patients with advanced/metastatic NSCLC, who are refractory to standard treatment, or for which no standard treatment is available.
  Interventions: Drug: HLX43
- Thymic carcinoma (Part 2 Dose Expansion) (Experimental): Patients with advanced/metastatic Thymic carcinoma, who are refractory to first line platinum based standard treatment.
  Interventions: Drug: HLX43
- NSCLC failed to standard and docetaxel treatment (Part 2 Dose Expansion) (Experimental): Patients with advanced/metastatic NSCLC, who are refractory to standard treatment and docetaxel.
  Interventions: Drug: HLX43
- Stage IIIB, IIIC, or IV NSCLC without any prior treatment (Part 2 Dose Expansion) (Experimental): Patients with stage IIIB, IIIC, or IV NSCLC that cannot be treated with surgery or radiotherapy, positive PD-L1 expression and no EGFR sensitizing mutation or ALK/ROS gene rearrangement, no previous systemic anti-tumor therapy for NSCLC.
  Interventions: Drug: HLX43; Drug: HLX10

INTERVENTIONS:
Drug: HLX43 — Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), until progressive disease (PD) without any clinical benefit, initiation of other anti-tumor therapies, death, intolerable toxicity, or withdraw the informed consent (whichever occurs first).
  Other Names: Anti-PD-L1 ADC
Drug: HLX10 — All participants will receive serplulimab (300 mg Q3W) via intravenous infusion (IV) until PD without clinical benefits, initiation of new anti-tumor therapy, death, intolerable toxicity, or withdrawal of informed consent (whichever occurs first), and serplulimab will be administered for up to 2 years (35 dosing cycles).
  Other Names: Serplulimab
  Arms: Stage IIIB, IIIC, or IV NSCLC without any prior treatment (Part 2 Dose Expansion)

SUMMARY:
This study is an open-label first-in-human phase I clinical study to evaluate the safety, tolerability, and pharmacokinetic characteristics of HLX43 in patients with advanced/metastatic solid tumors.

DETAILED DESCRIPTION:
This study is an open-label first-in-human phase I clinical study to evaluate the safety, tolerability , and pharmacokinetic characteristics of HLX43 with escalated doses in the treatment of patients with advanced/metastatic solid tumors.

In the phase Ia of this study, a 3 + 3 dose escalation method will be adopted, and the patients will be administered with HLX43 at different doses via intravenous infusion. The DLT observation period lasts for 3 weeks after the first administration of HLX43.

In phase Ib of this study, The Safety Review Committee will recommend dose groups for expansion based on the safety, efficacy and PK data of the dose escalation phase. The dose expansion part will include 4 cohorts: advanced/metastatic non-small cell lung cancer (NSCLC) patients with prior failed standard treatment or no standard treatment available, advanced/metastatic thymic carcinoma (TC) patients with prior failed first line platinum based standard treatment, advanced/metastatic NSCLC patients with prior failed standard treatment and docetaxel treatment, and stage IIIB, IIIC, or IV NSCLC patients who have not received any prior treatment with positive PD-L1 expression and no EGFR sensitizing mutation or ALK/ROS gene rearrangement.

ELIGIBILITY:
Inclusion Criteria:

1. Have a full understanding of the study content, process, and possible adverse reactions before the study, and sign the informed consent form (ICF); voluntarily participate in the study; be able to complete the study as per protocol requirements;
2. ≥ 18 years and ≤ 75 years at the time of signing the ICF, male or female;
3. In phase Ia, enroll patients with histologically or cytologically confirmed advanced/metastatic malignant solid tumors, who are refractory to standard treatment, or for which no standard treatment is available; In phase Ib Cohort 1: enroll patients with histologically or cytologically confirmed advanced/metastatic NSCLC, who are refractory to standard treatment, or for which no standard treatment is available (The standard treatment for squamous NSCLC is defined as platinum-containing chemotherapy combined with immune checkpoint inhibitor [ICI]. The standard treatment for non-squamous NSCLC with known EGFR mutations is defined as EGFR inhibitors and platinum-containing chemotherapy. The standard treatment for patients with non-squamous NSCLC without EGFR mutations is defined as platinum-containing chemotherapy combined with immune checkpoint inhibitor [ICI] therapy); Cohort 2: enroll patients with histologically or cytologically confirmed advanced/metastatic TC, who are refractory to first line platinum based standard treatment; Cohort 3: enroll patients with histologically or cytologically confirmed advanced/metastatic NSCLC, who are refractory to standard treatment and docetaxel treatment (The standard treatment for squamous NSCLC is defined as platinum-containing chemotherapy combined with immune checkpoint inhibitor [ICI]. The standard treatment for non-squamous NSCLC with known EGFR mutations is defined as EGFR inhibitors and platinum-containing chemotherapy. The standard treatment for patients with non-squamous NSCLC without EGFR mutations is defined as platinum-containing chemotherapy combined with immune checkpoint inhibitor [ICI] therapy); Cohort 4: enroll patients with histologically or cytologically confirmed stage IIIB, IIIC, or IV NSCLC that cannot be treated with surgery or radiotherapy; positive PD-L1 expression (PD-L1 positive is defined as TPS ≥ 1%; PD-L1 expression is subject to the central laboratory result) and no EGFR sensitizing mutation or ALK/ROS gene rearrangement; no previous systemic anti-tumor therapy for NSCLC (Patients who have received adjuvant or neoadjuvant therapy are allowed to be enrolled if the adjuvant/neoadjuvant therapy has been completed at least 6 months before the diagnosis of stage IIIB, IIIC, or IV NSCLC);
4. At least one measurable lesion as per RECIST 1.1 within 4 weeks prior to the first administration;
5. An ECOG performance status score of 0-1 within 7 days prior to the first administration;
6. Life expectancy > 3 months;
7. The following conditions must be met in terms of the time of the first administration of the investigational product: at least 28 days from the previous major surgery, medical device treatment, locoregional radiotherapy (except for palliative radiotherapy for bone lesions), cytotoxic chemotherapy, immunotherapy, or biological product therapy; at least 14 days from the previous small molecule targeted drug therapy and previous hormone therapy; at least 7 days from the administration of the traditional Chinese medicine for anti-tumor indications, or minor surgery; and recovery of treatment-induced AEs to grade ≤ 1 (CTCAE v5.0, except for alopecia);
8. Subjects who agree to provide archived tumor tissue specimens that meet the testing requirements (either from the most recent surgery or biopsy, preferably within 2 years) or agree to undergo a biopsy to collect tumor tissue for PD-L1 expression testing; Note: Formalin-fixed paraffin-embedded (FFPE) tumor samples (paraffin blocks or unstained sections, which must meet the quality control criteria for testing) collected from sites not receiving radiotherapy during the most recent surgery or biopsy at or after the diagnosis of malignant tumor and pathological reports of such specimens shall also be provided.
9. Adequate organ functions as confirmed by laboratory tests within 7 days prior to the first administration of the investigational product (no blood transfusions or treatment with granulocyte colony-stimulating factor within 14 days prior to the first administration).
10. For patients with hepatocellular carcinoma, Child-Pugh score must be A;
11. Male and female subjects with child-bearing potential must agree to use at least one highly effective contraception method during the study and within at least 6 months (at least 8 months for Japanese subjects) after the last administration of the investigational product; female subjects of childbearing age must have a negative pregnancy test within 7 days prior to enrollment.

Exclusion Criteria:

Subjects who meet any of the following criteria are not allowed to be enrolled:

1. Patients who have history of other malignant tumors within 2 years prior to the first administration, except for cured cervical carcinoma in situ or cutaneous basal cell carcinoma;
2. Patients who previously have immune-related adverse events (irAEs) ≥ grade 3 in immunotherapy;
3. Patients who have history of (non-infectious) interstitial lung disease (ILD) requiring steroids, or current ILD, or suspected ILD that cannot be ruled out by imaging at screening;
4. Subjects who are known to have anaphylaxis to protein preparations/monoclonal antibodies or are allergic to any component in the formulation of the investigational product;
5. Patients who have active systemic infectious diseases requiring intravenous antibiotics within 2 weeks prior to the first administration of the investigational product;
6. Subjects who have any poorly-controlled cardiovascular and cerebrovascular clinical symptoms or diseases, including but not limited to: (1) NYHA Class II or greater heart failure or left ventricular ejection fraction (LVEF) < 50%; (2) unstable angina pectoris; (3) myocardial infarction or cerebrovascular accident within 6 months (except for lacunar infarction, slight cerebral ischemia, or transient ischemic attack); (4) poorly controlled arrhythmia (including QTc intervals ≥ 450 ms for males and ≥ 470 ms for females) (QTc intervals are calculated by Fridericia's formula); (5) poorly-controlled hypertension (systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg after active treatment);
7. Patients who have been assessed as unsuitable for inclusion by the investigator, due to brain metastases, spinal cord compression, or cancerous meningitis with clinical symptoms, or uncontrolled brain or spinal cord metastases that have been evidenced; Note: Patients with asymptomatic or stable brain metastases, spinal cord compression, or cancerous meningitis as judged by the investigator are allowed to be enrolled;
8. Patients with known active or suspected autoimmune diseases. Those with autoimmune-related hypothyroidism and receiving thyroid hormone replacement therapy and those with type 1 diabetes mellitus controlled with insulin therapy are eligible to be enrolled;
9. Patients who have received systemic corticosteroids (prednisone > 10 mg/day or an equivalent dose of a similar drug) or other immunosuppressive agents within 14 days prior to the first administration; Except for the following circumstances: patients treated with topical, ocular, intra-articular, intranasal, and inhaled corticosteroids; those with short-term use of corticosteroids for prophylaxis if a contrast agent is used;
10. Patients who have used potent inhibitors or inducers of CYP2D6 or CYP3A within 2 weeks prior to the first administration;
11. Patients with active tuberculosis;
12. Patients who have history of immunodeficiency, including human immunodeficiency virus (HIV) infection or other acquired or congenital immunodeficiencies, or history of organ transplantation;
13. Patients with active HBV or HCV infection or HBV/HCV co-infection; Note: Patients who are HBsAg (+) and/or HBcAb (+) must undergo an HBV-DNA test and have a result of < 500 IU/mL, < 2500 copies/mL, or < ULN to be enrolled. Eligible subjects with detectable HBV-DNA must agree to receive anti-hepatitis B virus nucleoside treatment.

    Patients who are HCV antibody (+) must undergo an HCV-RNA test and have a result < ULN to be enrolled.

    Subjects with HBV/HCV co-infection shall be excluded (positive for HBsAg or HBcAb and positive for HCV antibody)
14. Patients who have received live vaccines within 28 days prior to the first administration;
15. Pregnant or lactating women (for Japanese subjects, pregnancy includes situations where the investigator believes that the subject may be pregnant, and lactating women can be enrolled in the study if breastfeeding is stopped, but breastfeeding cannot be resumed after receiving the study treatment);
16. Subjects who are not suitable for participating in this clinical study due to any clinical or laboratory abnormalities or other reasons as assessed by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
The Dose-Limiting Toxicity (DLT) of HLX43 within 21 days after the first Administration | From first dose to the end of Cycle 1 (each cycle is 3 weeks)
  DLT refers to the AEs that are determined to be related to the investigational product by the investigator, whose severity will affect the escalation of dose level. In this study, the DLT observation period lasts for 21 days after the first administration of HLX43.
Objective response rate (ORR) | approximately up to 24 months
  Percentage of participants with complete response (CR) and partial response (PR) based on investigator assessment.
The maximum tolerated dose (MTD) of HLX43 | From first dose to the end of Cycle 1 (each cycle is 3 weeks)
  The highest dose level, at which DLT is observed in no more than one of 6 evaluable patients, is defined as MTD of HLX43
RP2D | approximately up to 24 months
  The recommended phase 2 dose of HLX43

SECONDARY OUTCOMES:
Duration of response (DOR) | approximately up to 24 months.
  Length of time response continued based on investigator's assessment.
Progression-free survival (PFS) | approximately up to 24 months
  The PFS is defined as the time from the date of enrollment to the date of the first objective documentation of disease progression (as per RECIST v1.1) or death due to any cause,whichever occurred first.
Overall survival (OS) | approximately up to 24 months
  Time from the date of enrollment to the date of death for any cause.
Cmax | Up to 21 days after the first dose
  Maximum serum concentration (Cmax) of HLX43.
Tmax | Up to 21 days after the first dose
  Time to maximum serum concentration (Tmax) of HLX43.
T1/2 | Up to 21 days after the first dose
  Half-life (T1/2) of HLX43.
ADA (anti-drug antibody) | approximately up to 24 months
  Incidence and titer of ADA of HLX43.
Nab (neutralizing antibody) | approximately up to 24 months
  Incidence and titer of Nab of HLX43.
Number of subjects experiencing adverse events | Day 1 through 90 days after last dose.
  Frequency and seriousness of treatment emergent adverse events (TEAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, Dr., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Xiangya Hospital Central South University, Changsha, Hu'Nan

IPD SHARING:
Plan to Share IPD: No